CLINICAL TRIAL: NCT06921655
Title: Targeting prEssure-Muscle-index to Avoid Ventilatory Over-Assistance During Pressure
Brief Title: Targeting prEssure-Muscle-index to Avoid Ventilatory Over-Assistance During Pressure Support Ventilation
Acronym: TEMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Centre for Medical Sciences, Professor Giacomo Bellani, Università degli Studi di Trento
Organization: Università degli Studi di Trento (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TEMA
Record Dates: First submitted 2025-03-11; First posted 2025-04-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Acute Hypoxemic Respiratory Failure; Mechanical Ventilation Complication
Keywords: Pressure Support; Tidal Volume; Acute Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Randomized Cross-over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Pressure Support PMI=0 (Experimental): The PS level at which PMI is zeroed, meaning the patient's inspiratory effort contributes minimally to tidal volume
  Interventions: Procedure: Variation of Pressure Support Levels
- Pressure Support +2 (Experimental): Above PSPMI=0: +2 cmH₂O above PSPMI=0 (over-assistance zone).
  Interventions: Procedure: Variation of Pressure Support Levels
- Pressure Support +4 (Experimental): Above PSPMI=0: +4 cmH₂O above PSPMI=0 (over-assistance zone).
  Interventions: Procedure: Variation of Pressure Support Levels
- Pressure Support +6 (Experimental): Above PSPMI=0: +6 cmH₂O above PSPMI=0 (over-assistance zone).
  Interventions: Procedure: Variation of Pressure Support Levels
- Pressure Support -2 (Experimental): Below PSPMI=0: -2 cmH₂O below PSPMI=0 (under-assistance zone).
  Interventions: Procedure: Variation of Pressure Support Levels
- Pressure Support -4 (Experimental): - Below PSPMI=0: -4 cmH₂O below PSPMI=0 (under-assistance zone).
  Interventions: Procedure: Variation of Pressure Support Levels
- Pressure Support -6 (Experimental): - Below PSPMI=0: -6 cmH₂O below PSPMI=0 (under-assistance zone).
  Interventions: Procedure: Variation of Pressure Support Levels

INTERVENTIONS:
Procedure: Variation of Pressure Support Levels — Patients will undergo six randomized PS levels (+2, +4, +6 cmH₂O above and -2, -4, -6 cmH₂O below PSPMI=0).

SUMMARY:
The TEMA study (Targeting prEssure-Muscle-index to avoid ventilatory over-Assistance during pressure support ventilation) is a prospective, interventional crossover trial investigating the relationship between pressure support (PS) and tidal volume (Vt) in ICU patients with acute hypoxemic respiratory failure (AHRF) receiving pressure support ventilation (PSV). The study aims to assess whether the Pressure-Muscle Index (PMI)-a marker derived from the difference between plateau and peak inspiratory pressure-can help identify the optimal level of ventilatory assistance, preventing over-assistance and its associated complications such as diaphragm atrophy and patient self-inflicted lung injury (P-SILI). By exploring the sigmoidal relationship between PS and Vt, the study seeks to define a physiological threshold (PMI=0) that may serve as a personalized target for PSV titration.

DETAILED DESCRIPTION:
The TEMA study is a prospective, interventional crossover trial designed to explore the physiological relationship between levels of pressure support (PS) and tidal volume (Vt) in mechanically ventilated ICU patients diagnosed with acute hypoxemic respiratory failure (AHRF). The goal is to identify a pressure support threshold beyond which over-assistance occurs, leading to excessive tidal volumes and suppression of respiratory muscle activity.

The central hypothesis is that the PS-Vt curve follows a sigmoidal pattern: an initial plateau phase with stable Vt is followed by a steep, compliance-driven increase in Vt at higher PS levels. The Pressure-Muscle Index (PMI), calculated as the difference between plateau pressure (Pplat) and peak airway pressure (Ppeak) during an inspiratory occlusion, is used to define this inflection point (PMI=0), which marks the transition from physiologically appropriate to excessive assistance.

Study Design: The study is conducted at the ICU of Santa Chiara Hospital (Trento, Italy) and includes seven levels of pressure support modulation-three above and three below the identified PMI=0 point. At each level, key physiological variables such as Vt, respiratory rate (RR), minute ventilation, PMI, and patient-ventilator asynchrony index are recorded.

A second evaluation between days 4-6 post-enrollment is planned for patients who remain intubated, to assess whether the PS-Vt relationship evolves over time, reflecting changes in respiratory drive and mechanics during the ICU course.

Technical Aspects:

Measurements include respiratory system compliance, work of breathing (WOB), inspiratory effort, and occlusion-based indices.

PS levels are applied in randomized order to minimize bias. Clinical PSV settings are reinstated between steps to avoid carryover effects and ensure patient safety.

Analytical Approach: The primary outcome is to characterize the PS-Vt relationship and validate the use of PMI as a physiological marker of the optimal support threshold. Nonlinear regression models, including sigmoidal curve fitting, will be used to identify inflection points (c parameters) in the PS-Vt curve. A Monte Carlo simulation informed the sample size, targeting 36 patients to account for potential dropouts, ensuring >90% power to detect a meaningful breakpoint.

Multivariable models will adjust for potential confounders such as PaCO₂, sedation depth, BMI, and baseline compliance.

Expected Impact: If successful, the TEMA study will provide a new physiologically grounded framework for tailoring pressure support in assisted ventilation. By validating PMI as a real-time bedside tool, the study may support a more personalized approach to weaning and ventilation management, potentially improving outcomes such as duration of ventilation, weaning success, and ICU stay.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Mechanically ventilated in the ICU
3. Diagnosis of Acute Hypoxemic Respiratory Failure (AHRF)
4. Normocapnia or non-severe hypercapnia
5. Receiving Pressure Support Ventilation (PSV) for at least 24-72 hours
6. Presence of an arterial line for blood gas sampling

Exclusion Criteria:

1. Age < 18 years
2. Known neurological or neuromuscular disorders affecting diaphragm function
3. Chronic Obstructive Pulmonary Disease (COPD) or hypercapnic respiratory failure
4. Psychomotor agitation or inadequate sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2027-04-08 (Estimated); Study Completion 2027-04-08 (Estimated)

PRIMARY OUTCOMES:
Pressure Support-Tidal Volume (PS-Vt) Relationship | Up to 5 minutes after each PS level adjustment during the interventional phase (Day 1)
  The primary aim is to determine whether the PS-Vt curve exhibits a flat region (where tidal volume remains stable) before transitioning into a steep, compliance-dependent increase at higher PS levels. This transition point, identified as PSPMI=0, is hypothesized to represent the threshold for over-assistance.

SECONDARY OUTCOMES:
Validation of Pressure-Muscle Index (PMI) as an Over-Assistance Marker | Up to 5 minutes after each PS level adjustment during the interventional phase (Day 1) and during follow-up assessment on Days 4-6 (if patient remains intubated)
  PMI will be tested as a real-time bedside indicator for detecting over-assistance in PSV. The study will assess whether PMI=0 reliably corresponds to the threshold of over-assistance, characterized by a minimal patient contribution to Vt and a linear increase in Vt proportional to PS.
Impact of Respiratory Mechanics on PS-Vt Relationship | During the interventional phase on Day 1 and during follow-up assessment on Days 4-6 (if patient remains intubated)
  Evaluation of how respiratory compliance (Crs) influence the PS-Vt curve. The study will investigate individual variations in ventilatory response to PS.
Rate of Ineffective Efforts During Over-Assistance | Up to 5 minutes after each PS level adjustment during the interventional phase (Day 1) and during follow-up assessment on Days 4-6 (if patient remains intubated)
  Quantification of ineffective respiratory efforts (i.e., inspiratory efforts not followed by ventilator-triggered breaths) during PS levels exceeding the identified PSPMI=0 threshold.
Effect of Over-Assistance on Ventilatory Asynchronies | Up to 5 minutes after each PS level adjustment during the interventional phase (Day 1) and during follow-up assessment on Days 4-6 (if patient remains intubated)
  Measurement of the asynchrony index (percentage of breaths with any form of patient-ventilator asynchrony) at different levels of pressure support, particularly above PSPMI=0.
Weaning failure | Up to 100 months or until the of death from any cause, whichever came first.
  Defined as the inability to transition from PSV to unassisted breathing, requiring either reintubation, prolonged PSV dependence, or failure of a spontaneous breathing trial (SBT). The rate of weaning failure will be compared between patients receiving higher vs. lower levels of PSV support.
Duration of mechanical ventilation | From date of randomization until the date of extubation or date of death from any cause, whichever came first, assessed up to 100 months
  Total number of days on invasive mechanical ventilation (IMV), including both fully controlled and pressure-supported modes. The study will compare patients requiring different levels of PSV assistance.
ICU length of stay (LOS) | Up to 100 months or until the of death from any cause, whichever came first.
  Total duration (in days) of ICU admission, analyzing whether PSV settings influence prolonged ICU stays due to delayed weaning, respiratory complications, or ventilatory asynchronies
Hospital length of stay (LOS) | Up to 100 months or until the of death from any cause, whichever came first.
  Total number of days spent in the hospital from admission to discharge, evaluating whether PSV-related ventilatory strategies impact overall hospitalization duration and recovery time.
Impact of Respiratory Mechanics on PS-Vt Relationship | From the randomization to 5 minutes.
  Evaluation of how respiratory drive influence the PS-Vt curve. The study will investigate individual variations in ventilatory response to PS.
Impact of Respiratory Mechanics on PS-Vt Relationship | From the randomization to 5 minutes.
  Evaluation of how patient effort (Pmus) influence the PS-Vt curve. The study will investigate individual variations in ventilatory response to PS.
Spontaneous breathing failure | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Defined as the Number of Participants who fail transition from PCV to PSV.

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Chiara Hospital, Trento, Trentino-Alto Adige, Italy, Trento, Trento, Italy

IPD SHARING:
Plan to Share IPD: Undecided